CLINICAL TRIAL: NCT04259905
Title: Pink Warrior 2.0: Teleconference Support Group Toolkit for Breast Cancer Survivors
Brief Title: Pink Warrior 2: Teleconference-based Gaming Support
Acronym: PW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: M.D. Anderson Cancer Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-0040-02; 5P30AG024832 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-07 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Physical Activity
Keywords: active video game; telemedicine; cancer survivor; women's health; support group; survivorship; mhealth
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active video game teleconference support group (Experimental): Participants will attend enhanced support group meetings via zoom teleconferencing software. Support group meetings will include group play of active video games and discussion of survivorship topics. Participants will self-monitor physical activity using Fitbit wearable activity monitors and will receive a water bottle and tote bag.
  Interventions: Behavioral: Active video game teleconference support group
- Standard support group + pedometer (Active Comparator): Participants will attend standard in-person support groups currently offered by the UTMB Breast Health Center. They will also receive a standard pedometer and a water bottle and tote bag.
  Interventions: Behavioral: Standard support group + pedometer

INTERVENTIONS:
Behavioral: Active video game teleconference support group — 12 sessions of teleconferenced support group meetings, including active video game play + self-paced walking monitored by Fitbit wearable device
  Arms: Active video game teleconference support group
Behavioral: Standard support group + pedometer — 3 monthly sessions of in-person standard support group meetings + self-paced walking monitored by pedometer
  Arms: Standard support group + pedometer

SUMMARY:
Breast cancer survivors, from diagnosis until the end of life, go through many transitions. One major transition is the significant decrease of physical activity immediately after diagnosis. Despite the known benefits of physical activity-speeding recovery time and reduced cancer recurrence risk-only 1 in 3 survivors met physical activity recommendations of 150 minutes of moderate-intensity activity per week. Physical activity interventions have shown effectiveness in helping breast cancer survivors increase physical activity during treatment, but limited evidence-based physical activity interventions have been incorporated into the clinic and community. To address this limitation, the investigators are partnering with the UTMB breast cancer support group to conduct a 12-week physical activity intervention, Pink Warrior.

The goal of this study is to compare an intervention that uses active games versus an intervention uses pedometer to encourage physical activity such as walking within breast cancer survivors in active cancer treatment. The study will include breast cancer survivor between the ages of 18 - 70 whom currently gets less than 150 minutes of planned physical activity per week and received a breast cancer diagnosis within 0 to 6 months. Participants will be randomized to participate in the support group using the active video game-based physical activity intervention (Wii and Xbox active games) or to participate in the existing UTMB breast cancer support group with pedometers (Digi-Walker CW-700/701). The investigators hypothesize that by engaging in active video gaming, breast cancer survivors will be motivated to initiate and maintain physical activity during treatment. This will ultimately increase functional capacity and prevent functional disability in breast cancer survivors.

DETAILED DESCRIPTION:
Increasing and maintaining physical activity among female breast cancer (BC) survivors during treatment remains an unresolved problem in BC survivorship care. BC survivors, from diagnosis until the end of life, go through many transitions. One major transition is the significant decline of physical activity immediately after diagnosis. Despite the known benefits of physical activity-speeding recovery time and reduced cancer recurrence risk-less than 30% of survivors met physical activity recommendations. Physical activity interventions have shown effectiveness in helping BC survivors increase activity during treatment, but limited evidence-based activity interventions have been disseminated into the clinic and community. To address this limitation, we are partnering with the UTMB breast cancer support group to conduct a 12-week physical activity intervention, Pink Warrior, which will investigate the feasibility of implementing active video game-based physical activity intervention among BC survivors undergoing treatment within the support group setting. Participants (N = 60) will be randomized to participate in the support group using the active video game-based physical activity intervention or to participate in the existing UTMB breast cancer support group with pedometers. Our specific aims are:

Aim 1: Evaluate the feasibility and acceptability of active video game-based physical activity intervention among BC survivors undergoing treatment within the support group setting. Measures of feasibility will include weekly attendance records, number of completed home-based worksheets, number of participants completing the program activities, technological issues, and adverse events.

Aim 2: Compare the support group using the active video game-based physical activity intervention to the existing UTMB breast cancer support group with pedometer. Primary outcomes will be changes in physical activity. Secondary outcomes will be changes in physical function, dietary pattern, and quality of life.

Aim 3: Develop tools for implementation of the Pink Warrior intervention within the clinic and community settings. A trainer's manual for the Pink Warrior intervention will be developed and UTMB Breast Cancer Support Group facilitators will be trained by research staff to implement the program.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. Diagnosed with primary female breast cancer
3. 55 years to 79
4. Able to speak, read, and write in English
5. Able to travel to UTMB locations and/or MD Anderson Victory Lakes
6. Able to move arms and les as well as ambulate
7. Has a smartphone, tablet or computer and daily access to a reliable internet

Exclusion Criteria:

1. Pregnancy
2. Diagnosed dementia
3. Currently engage in 150 minutes or more of planned moderate intensity physical activity
4. Currently involved in another physical activity intervention

Ages: 55 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - The University of Texas Medical Branch, Galveston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.90 (8.03) | 62.60 (4.20) | 63.75 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Walking Physical Activity as Measured by Change in Daily Steps From Baseline to 14 Weeks
Description: Difference in mean of daily steps taken from Actigraph accelerometer worn for 7 day period from baseline assessment to 14 week assessment
Time Frame: Baseline to 14 weeks
Population: One person dropped out of the study shortly after randomization in the standard group and did not have a baseline step value
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer
Number analyzed (Participants) | 10 | 9
steps | -229.52 (1905.94) | 1570.17 (2355.59)
Statistical Analysis 1: Comparison: Standard Support Group + Pedometer; Test type: Superiority; Cohen's d = 0.85

2. Secondary Outcome: Quality of Life as Measured by the Change in FACT-B Scores From Baseline to 14 Weeks
Description: Quality of life score as measured by the Functional Assessment of Cancer Therapy-Breast measure at follow-up, scored for physical, social, emotional, functional, and breast well-being (here we report the total score of these subscales). The range for this scale is 0-123, with 0 indicating a better outcome.
Time Frame: Baseline to 14 weeks
Population: One person dropped out of the standard group shortly after randomization. An additional person in each group had missing values at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer
Number analyzed (Participants) | 9 | 8
units on a scale | 8.72 (10.07) | -1.69 (2.84)
Statistical Analysis 1: Comparison: Active Video Game Teleconference Support Group vs Standard Support Group + Pedometer; Test type: Superiority; Cohen's d = 1.29

3. Secondary Outcome: Physical Performance as Measured by the Change in Short Physical Performance Battery Scores From Baseline to 14 Weeks
Description: Difference in physical performance as measured by Short Physical Performance Battery from baseline to 14 weeks. The numbers reported here are the sum of scores from the subscales. The range for this measure is between 0-12, with lower scores indicating better outcomes.
Time Frame: Baseline to 14 weeks
Population: One person in the standard group dropped out of the study shortly after randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer
Number analyzed (Participants) | 10 | 9
units on a scale | 1.6 (1.17) | 0.44 (1.01)
Statistical Analysis 1: Comparison: Standard Support Group + Pedometer; Test type: Superiority; Cohen's d = 1.06

4. Other Pre Specified Outcome: Walking Skills in Daily Life
Description: Walking skills as measured by the Figure-of-8 Walk test
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Hand Grip Strength
Description: Flexor muscle strength of hand and forearm measured by dynamometer
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Physical Function as Measured by the Senior Fitness Test
Description: Physical function scores on six components: chair stands, arm curls, chair sit and reach, back scratch, 8 foot up and go, and 2 minute step in place test
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Body Weight in kg
Description: Mean body weight as measured by a calibrated scale in a cancer clinic setting
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Waist Circumference in cm
Description: Mean waist circumference as measured by Seca-203 measuring tape
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Dietary Pattern
Description: Dietary pattern change measured by the National Health and Nutrition Examination Survey (2009-10) measuring fruits, vegetables, dairy/calcium, added sugar, whole grains/fiber, red meat, and processed meat consumption within the past 30 days
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Self-reported Physical Activity Minutes
Description: Minutes of physical activity as self-reported using the Community Healthy Activities Model Program for Seniors questionnaire
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Self-reported Physical Function
Description: Physical function score as measured by the PROMIS cancer-specific instrument (PROMIS-CA Bank v1.1-Physical Function)
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Fatigue
Description: Fatigue score as measured by the PROMIS cancer-specific instrument (PROMIS-Ca Bank v1.1-Fatigue)
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exercise Motivation Measured as Autonomous Regulation
Description: Autonomous regulation as measured by the Behavioral Regulation in Exercise Questionnaire-2
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Psychological Feelings Related to Exercise
Description: Perceptions of autonomy, competence, and relatedness as measured by the Basic Psychological Needs in Exercise scale. 11 items on a 5-point Likert scale. Range: 1 (I do not agree at all) to 5 (I completely agree) for each of the constructs-autonomy (1-20), competence (1-20), and relatedness (1-15). The higher the score means more autonomy, more competence, and relatedness.
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Self-regulation: Exercise Goal-Setting (EGS) and Exercise Planning and Scheduling Scale (EPS)
Description: Goal-setting and planning measures, adapted from a published, untitled series of items created by Rovniak et al for evaluation of technology-mediated health promotion content. 10 EGS and 10 EPS items on a 5-point Likert scale. Range: 1 (does not describe) to 5 (describes completely) of the goal setting and planning strategies. The higher the score means more exercise goal-setting and planning behavior. (Rovniak et al. Annals of Behavioral Medicine, 2002, 24(2): 149-156.)
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Feasibility - Adherence
Description: Adherence as measured by number of participants who complete at least 80% of program activities
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Feasibility - Attrition
Description: Attrition as measured by percentage of people who drop out of the program
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Feasibility - Technological Issues
Description: Technological issues will be measured by counting the number of reported occurrences
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Feasibility - Adverse Events
Description: Adverse events will be measured by counting the number of occurrences
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Acceptability Scale
Description: Acceptability and satisfaction will be assessed via Vandelanotte questionnaire with 5-point scale responses, measures are adapted from a published, untitled series of items created by Vandelanotte et al for evaluation of technology-mediated health promotion content. Acceptability and feasibility of 3 components on a 5-point Likert scale-activity monitor (7-item), program team (6-item), and the program itself (15-item). Ranged: 1 (strongly disagree) to 5 (strongly agree). The higher the score means that it is more acceptable and feasible.
  (Vandelanotte, C. and I. De Bourdeaudhuij (2003). "Acceptability and feasibility of a computer-tailored physical activity intervention using stages of change: project FAITH." Health Educ Res 18(3): 304-317 and Vandelanotte, C., et al. (2004). "Acceptability and feasibility of an interactive computer-tailored fat intake intervention in Belgium." Health Promot Int 19(4): 463-470.)
Time Frame: Baseline to 14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: PI review of screening call logs, group session documentation, and data collection was used to systematically assess instances of adverse events.
Arm/Group | Active Video Game Teleconference Support Group | Standard Support Group + Pedometer
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Due to COVID-19 restrictions, we were unable to complete collection of Senior Fitness Test or hand grip measures. These were moved from secondary to other pre-specified outcomes. Other objective measures were collected via videoconference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT04259905/Prot_SAP_000.pdf